CLINICAL TRIAL: NCT06969014
Title: Treatment of Pulmonary Tumors Using Disposable Microwave Ablation Electrodes and a Microwave Ablation System Guided by Bronchoscopy: An Exploratory Study
Brief Title: Transbronchial MWA for Pulmonary Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Canyon Medical (Unknown)
Responsible Party: Principal Investigator, Jiayuan Sun, vice dean of the hospital, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS25007
Record Dates: First submitted 2025-04-23; First posted 2025-05-13 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Transbronchial MWA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transbronchial microwave ablation (Experimental)
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Device: Microwave ablation — Microwave ablation of lung tumors

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of transbronchial microwave ablation for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Pathologically diagnosed as primary peripheral lung cancer, preoperative staging suggested clinical staging as T1N0M0, stage IA (including new-onset lung cancer after surgery and multiple primary lung cancer). Or it is a metastatic lung tumor, the primary lesion has been completely resected, and the maximum diameter of the tumor is ≤3cm, the number of tumors requiring intervention is ≤3.
3. The lesion to be ablated has been evaluated as feasible for microwave ablation treatment under bronchoscopy guidance.
4. Agree to undergo transbronchial MWA as initial treatment after being assessed unsuitable for surgery and radiotherapy or refusing surgery and radiotherapy, and sign informed consent.

Exclusion Criteria:

1. Diffuse lesions in both lungs, for which ablation therapy is ineffective;
2. Preoperative evaluation within one month reveals the presence of intrathoracic lymph node metastasis or extrapulmonary metastasis (excluding cases where extrapulmonary metastasis has been locally controlled);
3. Contraindications to bronchoscopy, or inability to tolerate or comply with bronchoscopic procedures;
4. Severe hemorrhagic tendency, or uncorrectable coagulation disorders (PT > 18 seconds, PTA < 40%);
5. Platelet count < 70 × 10^9/L, or ongoing anticoagulant and/or antiplatelet therapy that has not been discontinued for more than one week prior to ablation (with the exception of prophylactic low-molecular-weight heparin use);
6. Severe pulmonary function impairment, with a maximal ventilatory volume < 40%;
7. Concurrent malignancies with widespread metastasis, with an expected survival of less than three months;
8. Poor overall condition (including widespread metastasis, severe infection, high fever), infectious or radiation-induced inflammation surrounding the lesion, significant cachexia, severe organ dysfunction, severe anemia, or nutritional and metabolic disturbances that cannot be corrected in the short term;
9. Eastern Cooperative Oncology Group (ECOG) performance status score > 2 ;
10. Lesions planned for ablation have received radiotherapy within the past six months;
11. Active hepatitis B, active hepatitis C, known human immunodeficiency virus (HIV) infection (HIV-1/2 antibody positive), or other active infections that may impact the patient's ability to undergo treatment as determined by the investigator;
12. History of epilepsy, psychiatric disorders, or cognitive impairments;
13. Patients with implanted cardiac pacemakers;
14. Patients wearing metal jewelry or clothing with metallic components;
15. Pregnant or lactating women, and individuals planning to conceive or become pregnant during the study period;
16. Participation in any other clinical trial within three months prior to signing the informed consent form (non-interventional studies excluded);
17. Any other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate of main lesion at 6 months post-procedure | 6 months
  6 months after ablation surgery, the proportion of patients with the main lesion maintained complete ablation among all evaluable patients who received transbronchial microwave ablation treatment.

SECONDARY OUTCOMES:
Complete ablation rate at 6 months, 12 months post-procedure (calculated in units of ablation lesions) | 12 months
  This refers to the proportion of completely ablated lesions in the total ablated lesions at 6 months and 12 months after transbronchial MWA.
Complete ablation rate at 6 months, and 12 months post-procedure (calculated in units of patients) | 12 months
  This refers to the proportion of patients with all treated lesions completely ablated in all patients who received transbronchial MWA at 6 months and 12 months after transbronchial MWA.
Progression-free survival rate at 12 months post-procedure | 12 months
  The proportion of patients who are progression-free (without disease progression or death from any cause) at 12 months post-procedure in the total evaluable patients who received transbronchial MWA.
Overall survival rate at 12 months post-procedure | 12 months
  The proportion of subjects who remain alive from the start of treatment until 1 year post-treatment.
Local progression-free survival rate at 6,12 months post-procedure | 12 months
  The proportion of subjects who remain local progression-free from the start of treatment until 6,12 months post-treatment.
Technical success rate | immediately after transbronchial MWA
  It is defined as the proportion of ablation treatment surgeries where the ablation instrument is successfully placed in the target lesion and the ablation instrument is successfully removed after the completion of the treatment procedure among all ablation treatment surgeries.
Safety evaluation of medical device use | immediately after transbronchial MWA
  Evaluate whether the microwave therapy device's microwave output is normal and whether the cooling circulation system is normal. Evaluate whether the water flow of the disposable microwave ablation electrode is smooth, whether the rod temperature is normal, whether there is tissue adhesion during ablation, and whether there is coolant leakage.
ECOG Score | 12 months
  The Eastern Cooperative Oncology Group (ECOG) scoring criteria were used to evaluate the physical performance status of subjects during the screening period, 7 days after treatment or before discharge, 1 month after treatment, 3 months after treatment, 6 months after treatment, and 12 months after treatment. A decrease in the score ≥1 before and after was defined as an improvement in performance status, an increase of ≥1 point was defined as a decrease in performance status, and no change in the score was stable.

OTHER OUTCOMES:
Safety of intervention | 12 months
  All adverse events were recorded and evaluated according to CTCAE v5.0 (if applicable), and the relevance to the device itself and the procedure was evaluated. The incidence of device-related and procedure-related adverse events and serious adverse events was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No